CLINICAL TRIAL: NCT03953482
Title: Evaluation of Medical Care and Patient's Knowledge About the Behavior to Take on Secondary Prevention of Anaphylaxis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: PREVANA
Record Dates: First submitted 2019-05-15; First posted 2019-05-16 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Anaphylaxis
MeSH Terms: conditions — Anaphylaxis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Anaphylaxis is a hypersensitivity reaction systemic, generalized, severe, life-threatening that may result from exposure to a triggering factor. The prevalence of anaphylaxis is 0.05 to 2% in the general population. Most reactions appear within 30 minutes after contact with the triggering factor and last up to 6 hours. The main triggering factors are: 1/food, 2/hymenopteran bites, 3/drugs. The main treatment is the early administration of adrenaline by Intramuscular route on medical prescription or by AAI (adrenaline auto-injector) associated with the exclusion of the allergen. Adrenaline treatment should be administered as soon as possible, a failure or delay in the use of adrenaline is a risk factor for death. Anaphylaxis is a chronic disease and the patient must be informed from the first episode about the risk of recurrence and the risk of death he is exposed to. Patient education is essential for the complete removal of the triggering factor, recognition of anaphylaxis symptoms and use of AAI. The risk of recurrence is high given the difficulty to completely eliminate the favourable factor (mainly food causes and hymenopteran bites): 1/3 of deaths from food anaphylaxis occur at home, and the peak mortality rate is between 10 and 30 years old. The diagnosis of anaphylaxis can be difficult because the symptomatology can be so varied. It is under-diagnosed, which leads to a lack of medical care and therefore an under-prescription of AAI. Some American studies identifying emergency room visits for anaphylaxis find that in less than 30% of cases there is a prescription for AAI, in less than 40% of advices about triggering factor's eviction and in less than 20% a guidance to an allergology consultation. In France, the HAS published in 2013 a procedure to be followed after the treatment of a suspected anaphylaxis: the patient's management must be diagnostic, therapeutic and educational. It must be systematically based on three axes:

* the prescription of AAI with an explanation of its use,
* the provision of written information on the mechanism and symptoms of anaphylaxis, attitude to be followed in event of an anaphylactic reaction, and need for eviction if the allergen has been identified,
* guidance to an allergology consultation.

Therapeutic education for anaphylactic patients is essential given the risk involved. In an American study, it was shown that only 60% of teens and young adults suffering from food allergies report having AAI systematically with them. Information and education is therefore essential for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age ≥ 18 years
* Francophone patient
* Patient not opposing his participation in the research protocol
* Patient with a history of an anaphylactic reaction

Exclusion Criteria:

* Patient under tutorship or curatorship
* Patient deprived of liberty
* Patient presenting an allergic reaction or an anaphylaxis
* For patients presenting to emergencies at Groupe Hospitalier Paris Saint-Joseph (GHPSJ) : Unstable health estate (gravity criteria hemodynamic, respiratory or neurological and any pathologies with a severity that do not allow the questionnaire to be answered).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with a history of an anaphylactic reaction
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2019-08-16 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient's medical management after a first episode of anaphylaxis | Day 0
  Percentage of patients who had management with:
  * an adrenaline auto-injector prescription (yes/no)
  * an eviction advice distribution (yes/no),
  * an allergology consultation (yes/no).

SECONDARY OUTCOMES:
Patient's knowledge of attitude to have with anaphylaxis | Day0
  Percentage of correct answers to the study-specific questionnaire related to knowledge of attitude to have with a new anaphylactic reaction.

CONTACTS AND LOCATIONS:
Overall Officials: Eloïse P TRABATTONI, MD, Study Director — Fondation Hôpital Saint-Joseph
Locations (2):
- France (2):
  - Maison de santé porte de Vanves, Paris
  - Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: Yes